CLINICAL TRIAL: NCT05274958
Title: A Comparison of the Effectiveness of Telepsychiatry With a Randomized Waitlist Control Utilizing Patient Reported Outcome Measures (PROMs)
Brief Title: Effectiveness of Telepsychiatry With Randomized Waitlist Control Utilizing Patient Reported Outcome Measures
Acronym: PROMs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Virginia Polytechnic Institute and State University (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-1426; UL1TR003015 (NIH)
Record Dates: First submitted 2022-02-16; First posted 2022-03-11 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: PROMs; Waitlist; Telemedicine; Mental Health Disorder; Psychiatric or Mood Diseases or Conditions
Keywords: Measurement-based Care
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Patients on a waitlist to see psychiatry will be enrolled then randomized to usual care or an intervention with monthly PROMs and an educational video
Who Masked: Outcomes Assessor
Masking Description: The intervention and data collection will take place before the patient sees the psychiatry clinician. The outcomes assessor will not be involved in the patient care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial PROM plus monthly PROM plus educational video (Experimental): These patients receive usual care plus monthly PROMs and educational video(s) while on the waitlist
  Interventions: Behavioral: Patient-rated outcome measures and educational videos
- Usual Care (No Intervention): Patients will complete the initial bundle of PROMs, then no further PROMs while they remain on the waitlist

INTERVENTIONS:
Behavioral: Patient-rated outcome measures and educational videos — PROMs are scales that are validated in behavioral health for tracking symptoms of depression, anxiety, and other conditions. They can be self-administered or given by a clinician. Mytonomy videos are short, educational videos about the patient's primary condition. All patients receive PROMs on entering our clinic. The difference in this intervention is those randomized to the active treatment will receive monthly PROMs and mytonomy video(s) until their appointment with the clinician. Usual care patients will only have PROMs at the intake and then at the appointment with their assigned clinician.
  Arms: Initial PROM plus monthly PROM plus educational video

SUMMARY:
The utilization of patient reported outcome measures (PROMs) during in-person care allows for on-going assessment of the severity of mental illness and patient outcomes across treatment. Additionally, it provides immediate feedback on the patient's psychiatric status to both the patient and practitioner. Carilion Clinic - Psychiatry & Behavioral Medicine ambulatory clinic implemented PROMs prior to the start of the COVID-19 (Coronavirus Disease 2019) pandemic and continues to utilize them as part of patient care. All new patients are asked to complete an initial PROM bundle of assessments 24 hours before their initial appointment, including the Brief Adjustment Scale, Patient Health Questionnaire, Generalized Anxiety Disorder survey, US Alcohol Use Disorder Identification Test, and Drug Assessment Screening Test. Automatic monthly reminders to complete the assessments continue after the first visit with the clinician. Over the last 2 years, research members of Carilion Clinic Psychiatry and Virginia Tech Psychology have been actively using PROM data to assess psychiatric health outcomes before and after the outbreak of COVID-19 in the United States. Initial results indicate that patients who received care via telepsychiatry not only did not experience worsening symptoms, but showed improvements in depression, anxiety and psychological functioning. However, without a control group of untreated patients to compare, the impact of telepsychiatry plus PROMs remains unclear. A waitlist control group design would allow investigators to compare patients receiving telepsychiatry and repeated completion of PROMs (current practice) to patients referred to psychiatry, but not receiving telepsychiatry treatment or completing PROMs during the same period. In this study, investigators plan to randomize individuals on the waitlist to one of two groups to assess the influence of time alone awaiting initial psychiatric clinician assessment (no intervention) versus minimal intervention using repeated PROMs and microlearning patient education videos while awaiting initial psychiatric clinician assessment. This kind of design allows assessment for the influence of time and the type of health service contact that replicates the basics of measurement-based psychiatric services (measurement of symptomology and well-being), but with none of the benefits of psychiatric supports, interventions, and techniques.

DETAILED DESCRIPTION:
Patient-reported outcome measures are a component of Measurement-Based Care (MBC) that involves collaboration between patient and clinician using structured evaluations of patient symptoms to inform behavioral health treatment and clinical decisions. In clinical settings, MBC has been found to improve outcomes and decrease dropout. Since patient-reported outcome measures can be performed by patients or clinicians, in session or out of session, and in-person or via telemedicine, their application is particularly pertinent during or after a crisis. The COVID-19 pandemic abruptly accelerated the transition to telehealth for many and necessitated alterations to traditional therapeutic means. PROMs are a tool that can improve the telehealth experience by strengthening patient-clinician relationships strained by the use of telemedicine, and allows for tracking of patient symptoms, which can be discussed and intervened upon in session.

Over the last 2 years, research members of Carilion Clinic Psychiatry and Virginia Tech Psychology departments have been actively using PROM data to assess psychiatric health outcomes before and after the outbreak of COVID-19 in the United States (IRB approved protocol 20-905). Initial results indicate that patients who received care via telepsychiatry not only did not experience worsening symptoms, but showed improvements in depression, anxiety and psychological functioning. However, without a control group of untreated patients to compare, the impact of telemedicine plus PROMs remains unclear. A wait-list control group design would allow investigators to compare participants receiving telemedicine and repeated completion of PROMs (current practice) to participants referred to psychiatry, but not receiving telemedicine treatment or completing PROMs during the same time period. Investigators propose randomizing wait-list individuals to one of two groups to assess the influence of time alone awaiting initial psychiatric clinician assessment (no intervention) versus minimal intervention using repeated PROMs and reviewing microlearning patient education videos while awaiting initial psychiatric clinician assessment. This kind of design allows assessment for the influence of time and the type of health service contact that replicates the basics of measurement-based psychiatric services (measurement of symptomology and well-being), but with none of the benefits of psychiatric supports, interventions, and techniques.

As of July 2021, 32 Carilion psychiatric clinicians are engaged in Owl Insights, an MBC vendor. Approximately 500 unique individuals complete monthly PROMs through this system as part of routine clinical care. The research group recently conducted analyses of nearly 900 ambulatory adult psychiatric patients in ambulatory psychiatry at Carilion Clinic (CC&PBM) engaging in PROMs via telepsychiatry and in-person modalities. PROM results of a patient cohort in clinical care prior to the onset of COVID-19 (November 2019) through March 2021 demonstrated that depression, anxiety and psychological functioning did not decline as hypothesized but statistically improved. Data also show that the engagement rates range from 33 to 74% depending on demographic factors, and completion rates were significantly different for diagnostic group and payor status of the patient. The standard goal for MBC utilization is 80%, while the department goal is to have all patients participate in PROM completion. The research group has also completed focus groups of psychiatric clinicians and staff with regards to Owl Insights and PROMs within the past year, identifying barriers and facilitators to its use and plan training implementation for improved adherence and satisfaction (summary of focus group data and training outline- included in grant application, IRB approved protocol 20-1065). Since March 2020, CC-P&BM has been engaging with patients via telephone and several telehealth platforms. Currently, ambulatory psychiatry uses AmWell (Amwell telemedicine) service, a telehealth platform that provides secure telemedicine visits between clinician and patient. The department has documented between 2100-2300 adult telemedicine sessions monthly and 200-700 in-person visits per month between June 2020 and June 2021.

CC-P&BM currently has a wait-list of over 300 adults referred for mental health evaluation and treatment. Access to psychiatric clinicians remains insufficient despite increasing numbers of providers in the local clinic and the mental health needs associated with the pandemic are rising. As a result, a clinical intake coordinator (Licensed Professional Counselor) began in the CC-P&BM ambulatory clinic September 2021. This coordinator will individually contact people on the wait-list for psychiatric care by phone as part of routine care, beginning with the referrals most remote in time. The coordinator will complete an intake assessment for each wait-list individual who wants a psychiatric referral. Prior to the initial intake assessment by the intake coordinator, wait-list individuals will receive a bundle of PROMs automatically (through Owl Insights) to complete. These measures include the Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder survey (GAD-7), Brief Adjustment Scale (BASE-6), Drug Assessment Screening Test (DAST-10), US Alcohol Use Disorder Identification Test (USAUDIT), Covid Event Checklist and the Adult Behavioral Health Screen (ABHS), all of which are currently used in routine ambulatory care. The intake coordinator will complete the intake assessment, noting the completion, and scores of, the PROMs. Scores of the PHQ-9, GAD-7 and BASE-6 will be utilized to triage the most severe referrals and move them up for a sooner appointment (the triage system of scores and Nurse-Practitioner vs Medical Doctor screening questions are attached to this application). Any concern about patient safety is also addressed immediately during this intake and is also noted in the materials attached to this application. Up to this point, all intake coordinator/referral interaction are part of routine care.

If eligible and capable of consent based on intake coordinator clinical judgement, individuals will then be randomized to participate to the no intervention group (completion of screening PROMs only during the intake coordinator assessment) or the minimal intervention group (intake coordinator assessment, including PROM screening and then prospective monthly PROM completion in addition to assigned microlearning patient education videos). Investigators will analyze changes in PROM scores for individuals engaged in both wait-list groups and compare results to their PROM scores at the initial provider telemedicine visit and over time (6 months post first provider assessment). Consent may be in-person with hard copy consent forms and signatures or through e-Consent either in-person or remotely.

The goals of this study are to (1) measure the symptomology and well-being of adult individuals on a waitlist group referred to CC-P&BM clinic from their initial referral to their initial psychiatric session with PROMs monthly versus only at entry to the waitlist and entry to clinic and (2) use PROMs to assess whether there is a difference in clinical symptomology and well-being for patients during tele-treatment with their practitioner compared to waitlist Individuals.

ELIGIBILITY:
Inclusion Criteria: A:

* all patients referred and see in an academic outpatient psychiatry clinic who wish to enroll

Exclusion Criteria:

* patients unable to engage in measurement-based care, such as those with dementia or other cognitive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia O'Brien, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Anita Kablinger, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalin ML, Garlow SJ, Thertus K, Peterson MJ. Rapid Implementation of Telehealth in Hospital Psychiatry in Response to COVID-19. Am J Psychiatry. 2020 Jul 1;177(7):636-637. doi: 10.1176/appi.ajp.2020.20040372. No abstract available. PMID 32605442
- [Background] Lambert MJ, Whipple JL, Kleinstauber M. Collecting and delivering progress feedback: A meta-analysis of routine outcome monitoring. Psychotherapy (Chic). 2018 Dec;55(4):520-537. doi: 10.1037/pst0000167. PMID 30335463
- [Background] Lewis CC, Boyd M, Puspitasari A, Navarro E, Howard J, Kassab H, Hoffman M, Scott K, Lyon A, Douglas S, Simon G, Kroenke K. Implementing Measurement-Based Care in Behavioral Health: A Review. JAMA Psychiatry. 2019 Mar 1;76(3):324-335. doi: 10.1001/jamapsychiatry.2018.3329. PMID 30566197
- [Background] Torous J, Wykes T. Opportunities From the Coronavirus Disease 2019 Pandemic for Transforming Psychiatric Care With Telehealth. JAMA Psychiatry. 2020 Dec 1;77(12):1205-1206. doi: 10.1001/jamapsychiatry.2020.1640. No abstract available. PMID 32391857
- [Result] Augusterfer EF, Mollica RF, Lavelle J. Leveraging Technology in Post-Disaster Settings: the Role of Digital Health/Telemental Health. Curr Psychiatry Rep. 2018 Aug 28;20(10):88. doi: 10.1007/s11920-018-0953-4. PMID 30155744
- [Result] Douglas S, Jensen-Doss A, Ordorica C, Comer JS. Strategies to enhance communication with telemental health measurement-based care (tMBC). Pract Innov (Wash D C). 2020 Jun;5(2):143-149. doi: 10.1037/pri0000119. PMID 34888414

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 286 people on the waitlist for ambulatory psychiatry were contacted for participation and assessed for eligibility. 138 were excluded: not meeting inclusion criteria, n=21 and declined to participate, n=117.
  N=148 agreed to participate
Groups:
- Initial PROM Plus Monthly PROM: These patients receive usual care plus monthly PROMs while on the waitlist
  Patient-rated outcome measures and educational videos: PROMs are scales that are validated in behavioral health for tracking symptoms of depression, anxiety, and other conditions. They can be self-administered or given by a clinician. All patients receive PROMs on entering our clinic. The difference in this intervention is those randomized to the active treatment will receive monthly PROMs until their appointment with the clinician. Usual care patients will only have PROMs at the intake and then at the appointment with their assigned clinician.
Period: Overall Study
Arm/Group | Initial PROM Plus Monthly PROM | Usual Care
Started | 70 | 78
Completed | 48 | 43
Not Completed | 22 | 35
Not completed — Only completed 1 set of PROMs | 22 | 35

BASELINE CHARACTERISTICS:
Groups:
- Initial PROM Plus Monthly PROM: These patients received usual care plus monthly PROMs while on the waitlist.
  Patient-rated outcome measures: PROMs are scales that are validated in behavioral health for tracking symptoms of depression, anxiety, and other conditions. They can be self-administered or given by a clinician. All patients receive PROMs on entering our clinic. The difference in this intervention is those randomized to the active treatment will receive monthly PROMs until their appointment with the clinician. Usual care patients will only have PROMs at the intake and then at the appointment with their assigned clinician.
- Usual Care: Patients completed the initial bundle of PROMs, then no further PROMs while they remained on the waitlist.
- Total: Total of all reporting groups
Arm/Group | Initial PROM Plus Monthly PROM | Usual Care | Total
Number analyzed (Participants) | 70 | 78 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (13) | 36 (12) | 36 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 54 | 106
  Male | 18 | 24 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 70 | 78 | 148
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 12 | 17
  White | 62 | 66 | 128
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
PHQ-9 score [Mean (Standard Deviation); unit: units on a scale] | 14 (6) | 14 (6) | 14 (6)
GAD-7 score [Mean (Standard Deviation); unit: units on a scale] | 13 (6) | 12 (5) | 13 (6)
BASE-6 score [Mean (Standard Deviation); unit: units on a scale] | 27 (9) | 28 (9) | 27 (9)
DAST-10 score [Mean (Standard Deviation); unit: units on a scale] | 1 (1) | 1 (2) | 1 (2)
USAUDIT [Mean (Standard Deviation); unit: units on a scale] | 5 (6) | 4 (4) | 5 (5)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Symptomatology of Patients on Waitlist Via Patient Health Questionnaire (PHQ-9)
Description: assess symptoms of patients on waiting list to see psychiatry from their initial referral to their initial psychiatric session. Score 0-27, higher is more severe depression.
Time Frame: 11 months
Population: Final PHQ-9 scores for each arm compared to baseline scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PROM Plus Monthly PROM: These patients receive usual care plus monthly PROMs while on the waitlist
  Patient-rated outcome measures: PROMs are scales that are validated in behavioral health for tracking symptoms of depression, anxiety, and other conditions. They can be self-administered or given by a clinician. All patients receive PROMs on entering our clinic. The difference in this intervention is those randomized to the active treatment will receive monthly PROMs until their appointment with the clinician. Usual care patients will only have PROMs at the intake and then at the appointment with their assigned clinician.
Arm/Group | PROM Plus Monthly PROM | Usual Care
Number analyzed (Participants) | 43 | 48
score on a scale
  Initial | 13.41 (6.18) | 13.48 (6.90)
  Final | 13.60 (6.80) | 13.00 (6.32)
Statistical Analysis 1: Comparison: PROM Plus Monthly PROM vs Usual Care; Patient measures for both groups were first summarized descriptively with means and standard deviations. To compare the two groups, a t-test was used; Test type: Superiority; p < 0.05, t-test, 2 sided

2. Primary Outcome: Measurement of Symptomatology of Patients on Waitlist Via Generalized Anxiety Disorder Survey (GAD-7)
Description: Assess symptoms of patients on waiting list to see psychiatry from their initial referral to their initial psychiatric session. Score 0-21, higher is more anxious.
Time Frame: 11 months
Population: Final GAD-7 scores for each arm compared to baseline scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PROM Plus Monthly PROM | Usual Care
Number analyzed (Participants) | 43 | 48
score on a scale
  Initial | 12.53 (5.76) | 12.42 (5.40)
  Final | 12.35 (5.99) | 11.54 (5.65)

3. Primary Outcome: Measurement of Symptomatology of Patients on Waitlist Via Brief Adjustment Scale (BASE-6)
Description: Assess symptoms of patients on waiting list to see psychiatry from their initial referral to their initial psychiatric session. Score 6-42, higher is poorer function.
Time Frame: 11 months
Population: Final BASE-6 scores for each arm compared to baseline scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PROM Plus Monthly PROM | Usual Care
Number analyzed (Participants) | 43 | 48
score on a scale
  Initial | 26.74 (9.23) | 27.10 (9.23)
  Final | 27.32 (9.24) | 25.47 (9.10)

4. Primary Outcome: Measurement of Symptomatology of Patients on Waitlist Via US Alcohol Use Disorder Identification Test (USAUDIT)
Description: assess symptoms of patients on waiting list to see psychiatry from their initial referral to their initial psychiatric session. Score 0-46, higher is greater alcohol use severity.
Time Frame: Baseline
Population: The USAUDIT was administered at baseline only; patients with primary or significant substance use disorders were referred to the addiction medicine service.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PROM Plus Monthly PROMs: Initial PROM plus monthly PROMS baseline
- Usual Care: Initial PROMs baseline
Arm/Group | PROM Plus Monthly PROMs | Usual Care
Number analyzed (Participants) | 70 | 78
score on a scale
  Female: number analyzed (Participants) | 52 | 54
  Female | 3.54 (4.07) | 3.52 (3.74)
  Male: number analyzed (Participants) | 18 | 24
  Male | 3.22 (3.56) | 5.83 (7.52)

5. Primary Outcome: Measurement of Symptomatology of Patients on Waitlist Via Drug Assessment Screening Test (DAST-10)
Description: Assess symptoms of patients on waiting list to see psychiatry from their initial referral to their initial psychiatric session. Score 0-10, higher indicates greater substance use.
Time Frame: Baseline
Population: DAST-10 was administered at baseline only; patients with primary or significant substance use disorders were referred to the addiction medicine service.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PROM Plus Monthly PROMs | Usual Care
Number analyzed (Participants) | 70 | 78
units on a scale | 0.90 (1.87) | 0.55 (1.05)

ADVERSE EVENTS:
Time Frame: Data was collected over an 11-month time frame.
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored/assessed, but none observed.
Arm/Group | Initial PROM Plus Monthly PROM | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/78
Other Adverse Events (participants affected / at risk) | 0/70 | 0/78

LIMITATIONS AND CAVEATS:
This study has several limitations. There was no control group who underwent psychiatric treatment without PROMs. PROM scores were not shared with patients in the waitlist groups, nor were they given education about what the scores meant clinically. Data was collected during the COVID-19 pandemic from a single adult academic clinic, and patients were predominantly white and female, limiting the generalizability of the results to other settings or populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT05274958/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT05274958/ICF_001.pdf